CLINICAL TRIAL: NCT02529514
Title: Usage of Baclofen for Sleep Improvement After Cardiac Surgery
Status: Suspended | Phase: Phase 4 | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Damien Wertz, MD, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Baclo-Sleep
Record Dates: First submitted 2015-06-04; First posted 2015-08-20 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Sleep
Keywords: Baclofen; Cardiac Surgery; Polysomnography; Intensive Care Units; Sleep
MeSH Terms: interventions — Baclofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Baclofen (Active Comparator): Baclofen 25 mg per os for 7 days at 10 pm every day
  Interventions: Drug: Baclofen
- Placebo (Placebo Comparator): Placebo per os for 7 days at 10 pm every day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baclofen — 25 mg for 7 days at 10 pm every day
  Arms: Baclofen
Drug: Placebo — Placebo for 7 days at 10 pm every day
  Arms: Placebo

SUMMARY:
Baclo-Sleep trial aims to investigate the effect of baclofen on sleep after scheduled cardiac surgery.

DETAILED DESCRIPTION:
This is a prospective randomized single-blind study involving patients adults admitted to the University Hospital of Liege for a scheduled heart surgery.

The study is based on the oral administration of baclofen (or placebo) the evening Bedrooms (10 pm). This administration begins the day before surgery and ends 5th day after. Sleep is evaluated by various questionnaires at baseline, during the protocol and the end. In addition, a 24 polysomnography is performed the day after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elective cardiac surgery

Exclusion Criteria:

* Haemodynamic instability
* Epilepsy
* Psychotic disturbances
* Acute / Chronic respiratory failure
* Morbid obesity (BMI > 45 kg/m2)
* Sleep apnea (treated)
* Severe hepatic or renal failure
* Patient refusal

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Polysomnography (quantity & quality of sleep) | Participants will be followed for the duration of hospital stay, an expected average of 10 days
  Sleep assessment by polysomnography

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Damas, Professor, Study Director — Soins intensifs généraux
Locations (1):
- Centre Hospitalier Universitaire de Liège, Liège, Liège, Belgium